CLINICAL TRIAL: NCT03444896
Title: The Efficacy and Neural Mechanism of Acupuncture Treatment in Older Adults With Subjective Cognitive Decline: a Randomized Controlled Trial
Brief Title: The Efficacy and Mechanism of Acupuncture Treatment in Patients With Subjective Cognitive Decline
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Ping Zhou, doctor, Beijing Hospital of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2017BL-061-03
Record Dates: First submitted 2018-02-04; First posted 2018-02-26 (Actual); Last update posted 2019-06-17 (Actual); Status verified 2019-06

CONDITIONS: Subjective Cognitive Decline; Subjective Cognitive Complaint

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture group (Experimental)
  Interventions: Device: Acupuncture group
- Sham acupuncture group (Placebo Comparator)
  Interventions: Device: Sham acupuncture group

INTERVENTIONS:
Device: Acupuncture group — Acupuncture needles were placed at acupoints Baihui (DU20), Shenting (DU24), Fengfu (DU16), Fengchi (GB20), Danzhong (RN17), Zhongwan (RN12), Qihai (RN6), Neiguan (PC6), Zusanli (ST36), Xuehai (SP10), Xinshu (BL15), Yixi (BL45), Tongli (HT5), and Zhaohai(KI6). Electrodes were attached the needle holders of the Baihui (DU20) and Shenting (DU24). The acupuncture needles are inserted through the adhesive pads and are retained for 20 minutes in every course. Treatment will be conducted over a period of 3 months, at a frequency of two times per week.
  Arms: Acupuncture group
Device: Sham acupuncture group — Sham acupoint (SA) 1 located in the midpoint of Shuaigu and Touwei. SA2 located in the midpoint of Touwei and Yangbai. SA3 located in the midpoint of Tianyou and Tianrong. SA4 located in 4 cun above umbilicus and 1 cun right of umbilical midline (UM). SA5 located in 2 cun below umbilicus and 1 cun right of UM. SA6 1 cun outside the point 1/4 of the line between Shenmen and Shaohai. SA7 located in 1 cun outside the midpoint of Shaohai and Tongli. SA8 located in 6 cun above mediosuperior border of the patella. SA9 located in 3 cun below the Yanglingquan and middle of the gallbladder and bladder channels. SA10 located in midpoint between Jiexi and Qiuxu. SA11 and SA12 located in 2 cun from the lower border of spinous process of fifth or sixth thoracic vertebra. Electrodes were attached the needle holders of the bilateral SA 2. Procedures, and other treatment settings were the same in the acupuncture group but with no skin penetration, electricity output, or needle manipulation for de qi.
  Arms: Sham acupuncture group

SUMMARY:
This study evaluates the efficacy and mechanism of acupuncture treatment in patients with subjective cognitive decline. Half of patients will receive acupuncture treatment for 12 weeks, while the other half will receive sham acupuncture treatment for 12 weeks .

ELIGIBILITY:
Inclusion Criteria:

1. Male and female adults aged 55-75;
2. Native Chinese speakers with right-handed and at least a primary school education;
3. Self-reported persistent memory decline, which was confirmed by caregivers;
4. Normal general cognitive function and not meeting the criterion of mild cognitive impairment, as defined by performance within the normal range on both measures within at least one cognitive domain or in each of the three cognitive domains sampled (adjusted for age and education);
5. No or minimal impairment in activities of daily living;

Exclusion Criteria:

1. Presence of positive neurologic history (e.g., traumatic brain injury, stroke, Parkinson's disease, multiple sclerosis, etc.) ;
2. treatments that would affect cognitive function;
3. Presence of significant psychiatric history (e.g., bipolar disorder, schizophrenia, etc.) and/or severe anxiety and depression;
4. Presence of serious heart, kidney, liver, gastrointestinal, infectious, endocrine disease or cancer;
5. History of alcohol or drug abuse/addiction in nearly two years;
6. Any contraindications for magnetic resonance imaging (MRI) scans (e.g., aneurysm clip pacemaker, etc.);
7. Significant visual and/or auditory impairment uncorrected by aids, and unable to perform neuropsychological evaluations;
8. Currently enrolled in another research study;
9. Received acupuncture treatment in the preceding month.

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-04-25 (Actual); Primary Completion 2020-01 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Change in cognitive function | Changes from baseline at 12 weeks
  A composite score will be computed by averaging z-scores from Animal Fluency Test, Digit Symbol Substitution Test, Trail-Making Test Parts A and B, Stroop Color Word Test C, Digit Span Test, Boston Naming Test, Clock Drawing Test and Auditory Verbal Learning Test delayed recall and delayed recognition.

SECONDARY OUTCOMES:
Neuroplasticity outcome | baseline and 12 weeks
  Neuroplasticity outcome changes are measured by structural MRI (including DTI), task functional MRI, resting state functional MRI and arterial spin labeling.

OTHER OUTCOMES:
The degree of complaint in cognitive decline | baseline and 12 weeks
  measured by Subjective Cognitive Decline Questionnaire.
The sleep quality | baseline and 12 weeks
  Measured by Pittsburgh Sleep Quality Index
The depressive symptoms | baseline and 12 weeks
  Measured by Geriatric depression scale
The face recognition ability and sense of direction | baseline and 12 weeks
  Measured by Face recognition questionnaire and Santa Barbara Sense of Direction scale

CONTACTS AND LOCATIONS:
Locations (1):
- School of Acupuncture-Moxibustion and Tuina, Beijing University of Chinese Medicine, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zhou H, Wang L, Wei XY, Lee CK, Wang ZY, Yan CQ, Liu CZ, Wang X, Shi GX. Brain Connectivity and Topological Reorganization of Multiple Functional Networks in Subjective Cognitive Decline After Acupuncture Intervention: A Secondary Analysis of a Randomized Controlled Trial. J Integr Neurosci. 2025 Nov 27;24(11):45003. doi: 10.31083/JIN45003. PMID 41351443
- [Derived] Wang L, Su XT, Yang NN, Wang QY, Yang JW, Liu CZ. Electroacupuncture improves cerebral blood flow in pMCAO rats during acute phase via promoting leptomeningeal collaterals. J Cereb Blood Flow Metab. 2025 Aug;45(8):1507-1518. doi: 10.1177/0271678X241270240. Epub 2025 Feb 26. PMID 40007441
- [Derived] Wang X, Zhou H, Yan CQ, Shi GX, Zhou P, Huo JW, Yang JW, Zhang YN, Wang L, Cao Y, Liu CZ. Cognitive and Hippocampal Changes in Older Adults With Subjective Cognitive Decline After Acupuncture Intervention. Am J Geriatr Psychiatry. 2024 Aug;32(8):1014-1027. doi: 10.1016/j.jagp.2024.03.001. Epub 2024 Mar 7. PMID 38521736
- [Derived] Yan CQ, Zhou P, Wang X, Tu JF, Hu SQ, Huo JW, Wang ZY, Shi GX, Zhang YN, Li JQ, Wang J, Liu CZ. Efficacy and neural mechanism of acupuncture treatment in older adults with subjective cognitive decline: study protocol for a randomised controlled clinical trial. BMJ Open. 2019 Oct 10;9(10):e028317. doi: 10.1136/bmjopen-2018-028317. PMID 31601583